CLINICAL TRIAL: NCT06268431
Title: Oxytocin Rest to Reduce Cesarean Delivery in Prolonged Labor: An Open-Label, Randomized Controlled Trial
Brief Title: Oxytocin Rest to Reduce Cesarean Delivery
Acronym: ORCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43084
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Prolonged Labor; Failed Induction; Labor Dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60-minute oxytocin rest (Experimental)
  Interventions: Other: Oxytocin rest
- Usual care with continuous oxytocin infusion (No Intervention)

INTERVENTIONS:
Other: Oxytocin rest — 60-minute oxytocin rest
  Other Names: pit rest
  Arms: 60-minute oxytocin rest

SUMMARY:
Prolonged labor is usually managed with continuous oxytocin infusion. "Oxytocin rest" has been proposed as a strategy to resolve protracted labor in patients who have received continuous oxytocin without progress. This strategy involves discontinuing oxytocin then restarting infusion after a period of time, under the theory that washout of the oxytocin receptor will strengthen uterine contractions to improve labor progress. "Oxytocin rest" is performed on labor and delivery units across the United States. Yet, there is no randomized or prospective data to support the practice.

The purpose of this study is to assess whether oxytocin rest of 60 minutes in patients with prolonged labor reduces risk for cesarean delivery.

DETAILED DESCRIPTION:
This open-label randomized trial of consenting pregnant people with prolonged latent labor aims to determine whether 60-minute oxytocin rest reduces risk for cesarean when compared to continuous oxytocin infusion. As secondary aims, this trial will also assess the impact of 60-minute oxytocin rest on: measures of the length of labor, risk for adverse maternal and neonatal outcomes, and measures of patient autonomy and sense of control.

The investigators will enroll 350 patients with singleton pregnancies at ≥36 weeks gestation with prolonged labor in the latent phase, defined as cervical dilation <6cm after ≥8 hours since rupture of membranes and on continuous oxytocin. Both nulliparous and multiparous individuals undergoing induction or augmentation of labor will be included. Patients with any contraindication to continuous oxytocin at randomization, or for whom cesarean section is anticipated at randomization will be excluded. Patients with prolonged rupture of membranes and patients with intraamniotic infection prior to randomization will also be excluded.

Using blocked randomization via computer-generated randomization scheme, subjects will be randomized with equal probability to 60-minute oxytocin rest or usual care with continuous oxytocin. Trial participants and their health care team will be aware of their assignment. Participants in the intervention group will undergo 60-minute oxytocin rest. With the permission of the clinical team, they will be able to break from continuous fetal monitoring to rest, shower, walk, or eat during this time. After 60 minutes, oxytocin will be restarted at 2 mU/min and subsequently increased by 2 mU/min every 30 minutes to a maximum dose of 30 mU/min or until adequate contractions are seen. Subjects in the control group will receive continuous oxytocin infusion, increased by 2 mU/min every 30 minutes to a maximum dose of 30 mU/min or until adequate contractions are noted.

The remainder of labor care will be at the discretion of the clinical team. Prior to hospital discharge, demographic and clinical data from each participant and their infant will be obtained via chart review.

The primary site for the trial will be ChristianaCare Health System.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Singleton gestation in vertex presentation
* ≥36 weeks gestation
* Prolonged latent labor, defined as cervical dilation <6cm after ≥8 hours since rupture of membranes and on continuous oxytocin

Exclusion Criteria:

* Not meeting the above criteria
* Any contraindication to continuous oxytocin at time of randomization
* Cesarean section anticipated by the clinical team at time of randomization (for any reason excepting labor dystocia)
* >18 hours between rupture of membranes and randomization
* Known intraamniotic infection at randomization
* Fetal demise
* Any contraindication to vaginal delivery
* Maternal eclampsia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Cesarean rate | At time of delivery
  Number of participants delivered by cesarean

SECONDARY OUTCOMES:
Time to delivery (hours) | From randomization to delivery
  defined as time from enrollment to delivery time, regardless of mode of delivery
Time to vaginal delivery (hours) | From randomization to delivery
  defined as time from enrollment to delivery time, for patients with vaginal delivery (cesarean delivery censored)
Time to active labor (hours) | From randomization to delivery
  defined as time from enrollment to first exam with cervical dilation ≥6cm (cesarean delivery at <6cm dilation censored)
Duration of active labor (hours) | From randomization to delivery
  defined as time from first exam with cervical dilation ≥6cm to delivery time (cesarean delivery censored)
Composite maternal adverse outcome | From date of delivery to date of hospital discharge for mother, expected average of 3 days
  to include operative vaginal delivery, obstetric anal sphincter injury, postpartum wound complications (wound cellulitis requiring antibiotics, wound reopened for fluid collection or infection, wound dehiscence), intraamniotic infection, postpartum endometritis, postpartum hemorrhage, deep vein thrombosis (DVT)/pulmonary embolism (PE), ICU admission, maternal death
Composite neonatal adverse outcome | From date of delivery to date of hospital discharge for neonate (or up to 28 days of life)
  to include NICU admission ≥48 hours, APGAR score at 5 minutes <7, cord pH <7.00, intubation and mechanical ventilation ≥12 hours, neonatal sepsis, hypoxic ischemic encephalopathy, stillbirth or neonatal death
Labor Agentry Scale score | From date of delivery to date of hospital discharge for mother, expected average of 3 days
  The LAS is a validated tool that captures patient perception of control over the labor process. It will be administered to all enrolled patients between 6 and 96 hours after delivery. The scale asks subjects to rate their agreement with multiple statements about the labor process from 1 (almost always) to 7 (rarely), with interpretation of ratings varying by statement.
Rate of intraamniotic infection (IAI) | From randomization to delivery
  defined as maternal temperature ≥ 38.0°C in the intrapartum period and initiation of antibiotics in the intrapartum period
Rate of postpartum endometritis | From date of delivery to date of hospital discharge for mother, expected average of 3 days
  defined as maternal temperature ≥ 38.0°C in the postpartum period AND initiation of antibiotics in the postpartum period
Rate of postpartum hemorrhage | From date of delivery to date of hospital discharge for mother, expected average of 3 days
  defined as quantitative blood loss ≥ 1000 mL (preferred) OR estimated blood loss ≥ 1000 mL (if QBL not performed or not available)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa C Logue, Principal Investigator — Christiana Care Health Services; Matthew K Hoffman, Principal Investigator — Christiana Care Health Services
Locations (1):
- ChristianaCare Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT06268431/Prot_SAP_000.pdf